CLINICAL TRIAL: NCT00987155
Title: Spinal Cord Injury: Endurance, Strength and Cardiac Function Induced by Efficient Training Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4.2007.2271
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Disease
Keywords: Functional electrical stimulation cycling; arm crank; wheelchair; ergometry; paraplegia; spinal cord injury; exercise testing
MeSH Terms: conditions — Cardiovascular Diseases; Paraplegia; Spinal Cord Injuries | interventions — Ergometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high intensity interval training (Experimental): 8 weeks of high intensity 4 times 4 interval training at 85-90% of peak heart rate during hybrid cycling
  Interventions: Device: Ergometry

INTERVENTIONS:
Device: Ergometry — MetamaxII Cortex ergospirometry system (Cortex Biophysik GmbH, Germany). Arm cycling ergometer (Ergomed 840L, Siemens, GermanyMonark, Sweden), Electrically braked wheelchair ergometer (VP 100, Handisoft France)
  Other Names: Sensor Medics Vmax Spectra 229 version 10. 1; ERGYS 2 Rehabilitation system; Lactate Pro LT-1710 Analyzer; Polar® accurex watch; Thigh cuffs Criticares NIBP with Riester Metpak manometer; Motionstim 8, Medel Electronics (isometric FES)

SUMMARY:
1. Measurements of peak oxygen uptake (VO2peak) during passive leg cycling (PLC) combined with arm crank ergometry (ACE), leg vascular occlusion (100mmHg above systolic BP) combined with ACE, and FES isometric contractions combined with ACE in spinal cord injured (SCI). All the above mentioned parameters will be compared to Functional Electrical Stimulated (FES) lower extremity cycling combined with ACE (FEShybrid). The hypothesis is that VO2peak is significantly higher during FES hybrid cycling when compared to peak and submaximal PLC, leg vascular occlusion and ACE. But the values for VO2peak during FES isometric contractions combined with ACE is not significantly different from FES hybrid cycling.
2. Comparison of sub-maximal and peak VO2 values during arm crank (ACE) and wheelchair ergometry (WCE) in persons with spinal cord injury. The hypothesis is that wheelchair propulsion due to higher energy expenditure show higher work output and VO2peak than ACE.
3. Does 6 weeks of maximal strength training improve SCI subjects performance during WCE? WCE after 6 weeks maximal strength training is less strenuous owing to better work economy/ efficiency.
4. Effect from aerobic high intensity hybrid training on stroke volume (SV) and VO2peak in spinal cord injured men.

8 weeks of high intensity 4 times 4 interval training at 85-90% of peak heart rate during hybrid cycling. Hypothesis; VO2peak and SV will be significantly increased from training.

ELIGIBILITY:
Inclusion Criteria:

* Paraplegia, sensorimotor complete injury AIS A to motor complete, sensory incomplete AIS B. Chronic neurological state with stabile spontaneous recovery compared to baseline AIS. At least year since injury.
* Be able to tolerate direct current stimulation in the means of FES
* Living in Health region IV and V, Norway.

Exclusion Criteria:

* Pacemaker (demand type)
* Known cancer
* Known pregnancy
* Severe autonomic dysreflexia
* Gross contractures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | 2 years

SECONDARY OUTCOMES:
Blood lactate | 2 years
Blood Pressure | 2 years
Perceived Exertion | 2 years
Generated power (W) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Leivseth, Professor MD, Principal Investigator — National Taiwan Normal University; Gisle Meyer, Study Director — St. Olavs Hospital; Lars Jacob Stovner, Professor, Study Director — National Taiwan Normal University; Jan Hoff, Professor, Principal Investigator — National Taiwan Normal University; Berit Brurok, MSc, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olav University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Torhaug T, Brurok B, Hoff J, Helgerud J, Leivseth G. Arm Crank and Wheelchair Ergometry Produce Similar Peak Oxygen Uptake but Different Work Economy Values in Individuals with Spinal Cord Injury. Biomed Res Int. 2016;2016:5481843. doi: 10.1155/2016/5481843. Epub 2016 Apr 10. PMID 27144169